CLINICAL TRIAL: NCT07017829
Title: A Phase II Trial of GT103 in Combination With Pembrolizumab in STK11 Mutant Non-Small Cell Lung Cancer (NSCLC)
Brief Title: GT103 in Combination With Pembrolizumab for the Treatment of Advanced or Metastatic STK11 Mutant Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-4003224; NCI-2024-08947 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-4003224 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Advanced Lung Non-Small Cell Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Stage III Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (GT103, pembrolizumab) (Experimental): Patients receive GT103 IV over 60 minutes and pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO at baseline, MRI at baseline and as clinically indicated, and CT and blood sample collection throughout the study. Patients may also undergo biopsy throughout the study.
  Interventions: Biological: Anti-CFH Monoclonal Antibody GT103; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Anti-CFH Monoclonal Antibody GT103 — Given IV
  Other Names: GT 103; GT-103; GT103
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475

SUMMARY:
This phase II trial tests how well GT103 in combination with pembrolizumab works in treating patients with STK11 mutant non-small cell lung cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic). GT103 is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. GT103 targets the tumor cell-protein complement factor H found on some cancer cells and may provide specific anti-tumor activity that may help block the formation of growths that may become cancer. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving GT103 in combination with pembrolizumab may kill more cancer cells and improve outcomes in patients with advanced or metastatic STK11 mutant non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the 6-month (24 week) progression-free survival (PFS) rate of anti-CFH monoclonal antibody GT103 (GT103) in combination with pembrolizumab in patients with advanced/metastatic STK11 mutant non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To evaluate secondary efficacy endpoints (i.e., investigator-assessed objective response rate, 12-month survival rate, overall survival, duration of response, and disease control rate) of GT103 in combination with pembrolizumab in patients with advanced/metastatic STK11 mutant NSCLC.

II. To evaluate the safety and tolerability of GT103 in combination with pembrolizumab in advanced/metastatic STK11 mutant NSCLC.

EXPLORATORY OBJECTIVES:

I. To evaluate the effects of GT103 in combination with pembrolizumab on the tumor microenvironment.

II. To explore study tissue and blood-based biomarkers as potential predictors of treatment efficacy.

OUTLINE:

Patients receive GT103 intravenously (IV) over 60 minutes and pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography (ECHO) at baseline, magnetic resonance imaging (MRI) at baseline and as clinically indicated, and computed tomography (CT) and blood sample collection throughout the study. Patients may also undergo biopsy throughout the study.

After completion of study treatment, patients are followed up every 30 days for 120 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 at the time of study treatment initiation.
* Have pathologically confirmed diagnosis of STK11 mutant NSCLC. STK11 mutation will be based on subject's local clinically accredited laboratory testing (Clinical Laboratory Improvement Amendments [CLIA]-certified) using deoxyribonucleic acid (DNA) sequencing test.
* Must have progressed on a pembrolizumab containing regimen and eligible for continuing pembrolizumab post-progression as determined by treating physician.
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L.
* Platelets ≥ 100 x 10^9/L.
* Hemoglobin ≥ 9 g/dL.
* Estimated glomerular filtration rate (GFR) (measured or calculated with Cockroft and Gault formula) > 45mL/min.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN) (ALT and AST ≤ 5 x ULN is acceptable if liver metastases are present).
* Total bilirubin ≤ 1.5 x ULN. For patients with well documented Gilbert's syndrome, total bilirubin ≤ 3 x ULN with direct bilirubin within normal range.
* Troponin-I ≤ ULN and B-type natriuretic peptide test (BNP) < 200 pg/mL.
* Left ventricular ejection fraction (LVEF) ≥ lower limit of normal (LLN) (institutional limit).
* Patients must have measurable disease as defined in Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.
* Participant agrees to provide blood samples at the start of treatment and at multiple times during the study. Participant agrees to provide tumor biopsy tissue or have adequate archival formalin-fixed paraffin-embedded (FFPE) tissue available.

Exclusion Criteria:

* Receipt of anticancer chemotherapy within 4 weeks before the first administration of study drug.
* Prior radiotherapy or gamma knife within 2 weeks of study treatment for non-brain metastasis. Subjects must have recovered from all radiation related toxicities.
* Active/untreated brain metastasis. Whole brain radiation or gamma knife radiosurgery performed less than 4 weeks prior to first administration of study drug. Previously treated brain metastasis allowed as long as not requiring steroids and stable on imaging at least 4 weeks after completing radiation therapy.
* Leptomeningeal involvement regardless of treatment status.
* Tumor with oncogenic mutation based on standard of care broad genomic profiling in EGFR, ALK, ROS1, RET, MET, or NTRK genes.
* History of autoimmune disorder, with exception of patients with vitiligo or endocrine-related autoimmune conditions receiving appropriate hormonal supplementation who are eligible. Systemic use of immunosuppressant drugs such as steroids (except as hormone replacement therapy or short-course supportive medication such as chemotherapy or drug allergy, etc.), azathioprine, tacrolimus, cyclosporine, etc. within 4 weeks before the first administration of study drug.
* Currently receiving or has received systemic corticosteroids within 4 weeks prior to starting study drug for management of brain metastases, or who have not fully recovered from side effects of such treatment. Steroids for endocrine replacement or receipt of short-course of steroids during the preceding 4 week period as supportive medication such as for drug allergy, anti-emetic, etc. is allowed.
* Had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered major surgery) resulting from a prior surgery.
* Has known immunosuppressive disease (e.g., HIV, AIDS or other immune depressing disease). Testing is not mandatory.
* Active, clinically serious infections or other serious uncontrolled medical conditions.
* Patient has known hypersensitivity to the components of the study drugs or any analogs.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator, including, but not limited to:

  * Myocardial infarction or arterial thromboembolic events within 6 months prior to baseline or severe or unstable angina, New York Heart Association (NYHA) Class III or IV disease.
  * History of documented congestive heart failure (New York Heart Association functional classification III or IV) within 6 months prior to baseline.
  * Uncontrolled hypertension (systolic blood pressure [SBP] > 160/diastolic blood pressure [DBP] > 100 despite medical intervention).
  * History of myocarditis of any etiology.
  * History of ventricular arrhythmias.
* Patients diagnosed with an invasive cancer within 2 years prior to starting protocol therapy with the following exceptions: non-melanoma skin cancers, in-situ cancers, and prostate cancer Gleason ≤ 6 (under surveillance or treated), early-stage node-negative estrogen receptor positive (ER+)/progesterone receptor positive (PR+) breast cancer with Oncotype Dx score < 25 not taking adjuvant hormonal therapy.
* Pregnant or nursing female participants.
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug.
* Unwilling or unable to follow protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Between study registration and documentation of disease progression or death, whichever is observed first, assessed up to 6 months (24 weeks)
  Will be summarized using standard Kaplan-Meier methods, where estimates will be obtained with 90% confidence intervals.

SECONDARY OUTCOMES:
Objective response rate | Up to 4 years
  Will be defined by the Response Evaluation Criteria in Solid Tumors version 1.1. Will be estimated using 90% credible regions obtained by Jeffrey's prior method.
Overall survival | Between registration and death from any cause, assessed up to 4 years
  Will be assessed using standard Kaplan-Meier methods, where estimates will be obtained with 90% confidence intervals.
Duration of response | From the first documented objective response until the first documented disease progression or death due to any cause, assessed up to 4 years
  Will be summarized using standard Kaplan-Meier methods, where estimates will be obtained with 90% confidence intervals.
Disease control rate | From the first dose of study drug until the first documentation of disease progression or death, assessed up to 4 years
  Will be defined as the proportion of patients with a best overall response of confirmed complete response, confirmed partial response, or stable disease ≥ 12 weeks. The best response status will be summarized using frequencies and relative frequencies.
Incidence of adverse events | Up to 120 days after end of treatment
  Toxicities and adverse events will be assessed per Common Terminology Criteria for Adverse Events version 5.0. Will be summarized by attribution and grade using frequencies and relative frequencies.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin H Yau, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States